CLINICAL TRIAL: NCT07003841
Title: Multicenter, Randomized, Controlled, Prospective, Confirmatory Study to Evaluate the Clinical Efficacy of Augmented Reality (AR)-Based Breast Cancer Medical Imaging Solution (SKIA-Breast) Localization Method in Breast Cancer Patients Confidential Statement
Brief Title: Evaluation of Clinical Efficacy of Augmented Reality (AR)-Based Breast Cancer Medical Imaging Solution (SKIA-Breast) Localization Method in Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SKIA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S_SKIAB_P02
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Navigation Systems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigational device and the control device used in this clinical trial have distinctly different appearances, making it impossible to maintain blinding of the investigators and participants; therefore, the trial will be conducted with blinding of an independent evaluator only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Skin Marking Group (Active Comparator): Mastectomy will be performed after applying the ultrasound skin marking method
  Interventions: Device: General ultrasound imaging system
- AR-based Imaging Group (Experimental): Mastectomy will be performed after applying the localization method using the augmented reality-based medical imaging solution
  Interventions: Device: Surgical navigation system with stereotactic guidance

INTERVENTIONS:
Device: Surgical navigation system with stereotactic guidance — This investigational medical software device utilizes CT imaging data to project the scanned anatomy onto the patient's body, enabling augmented reality-based visualization of the lesion site before surgery
  Other Names: SKIA-Breast
  Arms: AR-based Imaging Group
Device: General ultrasound imaging system — A general diagnostic ultrasound imaging device that transmits ultrasound energy to the lesion for diagnostic purposes and visualizes the reflected signals. It supports various types of transducers and associated application software packages used for acquiring, displaying, and analyzing ultrasound data.
  Arms: Ultrasound Skin Marking Group

SUMMARY:
This clinical trial aims to evaluate whether an augmented reality (AR)-based medical imaging solution (SKIA-Breast) is non-inferior to conventional ultrasound-guided skin marking in guiding breast-conserving surgery in female patients with breast cancer. Participants will be randomly assigned in a 1:1 ratio to either the AR-based group or the conventional group. All participants will undergo breast-conserving surgery according to their assigned method. The primary outcome is the negative margin resection rate evaluated by histopathological examination. The secondary outcome is the re-excision rate due to positive margins assessed by histopathological examination.

DETAILED DESCRIPTION:
1. Background With the increasing incidence of early breast cancer due to advancements in diagnostic imaging and screening, breast-conserving surgery (BCS) has become more common, offering improved patient satisfaction and quality of life. Accurate lesion localization is critical for successful BCS. While several localization techniques exist, no single method is widely standardized. Augmented reality (AR) presents a promising non-invasive alternative, enabling real-time visual projection of lesion and lymph node positions onto the skin, potentially improving surgical accuracy and addressing limitations of conventional methods.
2. Purpose This study aims to evaluate the clinical efficacy of an AR-based medical imaging localization method (SKIA-Breast) compared to conventional ultrasound-guided skin marking in patients diagnosed with breast cancer who require breast-conserving surgery.
3. Procedure This multicenter, randomized, controlled clinical trial will assess whether the AR-based medical imaging solution (SKIA-Breast) is non-inferior to conventional ultrasound-guided skin marking in guiding breast-conserving surgery. Female patients with breast cancer will be randomly assigned in a 1:1 ratio to either the AR-based group or the conventional group. All participants will undergo breast-conserving surgery according to their assigned method.

The primary outcome is the negative margin resection rate, evaluated by histopathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be enrolled only when all the inclusion criteria are fully met.

  1. Subjects who aged 19 to 80 years diagnosed with breast cancer through biopsy.
  2. Subjects diagnosed with breast cancer who had both MRI and CT and ultrasound scans.
  3. Patients diagnosed with breast cancer who are scheduled to undergo breast-conserving surgery, have not received neoadjuvant chemotherapy, and show no evidence of metastasis to other organs.
  4. Tumor size criteria on ultrasound: : 5 mm ≤ tumor size ≤ 30 mm
  5. Subjects whose biopsy pathology results are Invasive carcinoma.
  6. Subjects who have a single lesion.
  7. Subjects who have received a full explanation of the clinical trial fully understand its details, voluntarily decide to participate, and provide written informed consent.

Exclusion Criteria:

* Subjects will be excluded from enrollment if they meet any of the exclusion criteria.

  1. Subjects prohibited from both MRI, CT and Ultrasound scans.
  2. Subjects with no lesions visible on CT.
  3. Pregnant or lactating(i.e., breastfeeding) subjects.
  4. Subjects who are biologically male.
  5. Subjects with breast cancer who received neoadjuvant chemotherapy or who have metastasized to other organs
  6. Subjects whose biopsy pathology results are Invasive lobular carcinoma
  7. Subjects deemed unsuitable for the study according to judgment of the investigator

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Negative margin resection rate | within 4week after biopsy
  Each subject will have one surgical margin evaluated, with an independent pathologist determining margin status (negative or positive) based on the permanent postoperative pathology specimen. Measurements of the margin are taken in the medial, lateral, superior, and inferior directions in millimeters, with conservative rounding applied to decimal values.

SECONDARY OUTCOMES:
re-excision rate | within 4week after biopsy
  Re-excision rate due to positive margins assessed by histopathological examination
margin assessment | within 4week after biopsy
  In breast resections performed after the application of the investigational medical device, pathological assessment of the resection margins will be conducted by an independent evaluator (pathologist). Only the lateral, medial, superior, and inferior directions will be recorded, while the deep and superficial margins will be excluded.
  For analysis, the minimum value among the four recorded margins will be selected and classified into the following six categories:
  1. Less than 2 mm
  2. 2 mm to less than 5 mm
  3. 5 mm to less than 10 mm
  4. 10 mm to less than 20 mm
  5. 20 mm to less than 30 mm
  6. 30 mm or greater
Tumor-to-gross area ratio of excised tissue | within 4week after biopsy
  Tumor-to-gross area ratio of excised tissue (excluding thickness) assessed by histopathology.
  Calculation formula: (Tumor surface area / Gross (tumor + margin) surface area) × 100 (%)
User satisfaction | on the day of biopsy
  User satisfaction is assessed in the investigator's survey covering usability, safety, overall satisfaction, and reusability. This satisfaction is measured using a 5-point Likert scale, where higher scores indicate greater satisfaction following the application of the investigational medical device.

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Ewha Womans University Medical Center, Seoul, Gangseo-gu
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Yonsei University Health System, Severance Hospital, Seoul, Seodaemun-gu

IPD SHARING:
Plan to Share IPD: No